CLINICAL TRIAL: NCT03013465
Title: Daily Consumption of Well-Cooked Broccoli May Affect Glucosinolate Metabolites and Inflammatory Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Craig Charron, Research Molecular Biologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HS55
Record Dates: First submitted 2016-12-19; First posted 2017-01-06 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Diet (Other): Participants will receive a controlled diet (base diet), typical of an American diet, with 0 g/day of broccoli (control).
  Interventions: Other: Control Diet
- Brassica Diet (Active Comparator): Participants will receive a controlled diet with 100 g of broccoli at both breakfast and dinner daily.
  Interventions: Other: Base Diet with Broccoli

INTERVENTIONS:
Other: Control Diet — Participants will receive a controlled diet with 0 g/d of broccoli. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Other Names: Base Diet
  Arms: Control Diet
Other: Base Diet with Broccoli — Participants will receive a controlled diet with 100 g of broccoli at both breakfast and dinner daily. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Arms: Brassica Diet

SUMMARY:
The objectives of the study are 1) to determine the influence of daily consumption of well-cooked broccoli on plasma and urinary glucosinolate metabolites, and 2) to determine inflammatory marker changes consistent with decreased cancer risk.

DETAILED DESCRIPTION:
Consumption of Brassica vegetables is inversely associated with incidence of several cancers, including cancer of the lung, stomach, liver, colon, rectum, breast, endometrium, and ovaries. Brassica vegetables are a good source of many nutrients, but the unique characteristic of Brassicas (Broccoli in particular) is their rich content of glucosinolates. Glucosinolates are sulfur-containing compounds that are converted to isothiocyanates (ITC) by an enzyme in the plant called myrosinase, which is released when the vesicles containing myrosinase are ruptured by chewing or cutting. The isothiocyanates are considered to be the active agent for cancer prevention. Some of the mechanisms by which isothiocyanates likely inhibit cancer include modulation of cytochrome P450 enzymes, induction of phase II enzymes, and apoptosis.

The aim of this study is to investigate how daily consumption of broccoli with myrosinase inactivated by cooking influences glucosinolate metabolism and absorption, and consequent regulation of inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Non tobacco user
* Cancer Free
* Not currently taking glucosinolate/isothiocyanate containing supplements

Exclusion Criteria:

* Type 2 diabetes requiring the use of diabetes pills, insulin, or non-insulin shots
* Use of blood-thinning medications such as Coumadin (warfarin), Dicumarol, or Miradon (anisinidione)
* History of bariatric surgery or nutrient malabsorption disease
* Pregnant, lactating, or intending to become pregnant during the study period
* Crohn's disease or diverticulitis
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
The change in glucosinolate metabolites will be measured in blood plasma and urine | At end of diet period 1 (week 3) and at the end of diet period 2 (week 12)
  To track the change of endogenous broccoli isothiocyanates in this crossover study, glucosinolate metabolites will be measured in both blood plasma and urine

SECONDARY OUTCOMES:
Body composition will be determined by dual energy x-ray absorptiometry (DEXA) | Day 0, just prior to beginning the controlled diet
  Determine fat, lean, and bone mineral mass, and visceral fat deposition in our subjects
The ability of fecal microbiota to metabolize glucosinolates will be determined | once per week during diet periods 1 and 2 (weeks 1, 2, 3, 10, 11, and 12)
  Fecal samples will be presented with glucoraphanin to determine the ability of fecal microbes to metabolize it
Fecal microbiota will be analyzed for microbial DNA | once at the beginning and end of diet periods 1 and 2 (weeks 1, 3, 10, and 12)
  Fecal microbial communities will be determined using DNA extracted from fecal samples
Markers of gut health will be analyzed in blood | once in the third week of diet periods 1 and 2 (weeks 3 and 12)
  Zonulin in blood serum will be measured by ELISA
Markers of inflammation will be measured in blood | at end of diet period 1 (week 3) and at end of diet period 2 (week 12)
  Cytokines and acute phase proteins will be measured in blood

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charron CS, Vinyard BT, Jeffery EH, Ross SA, Seifried HE, Novotny JA. BMI Is Associated With Increased Plasma and Urine Appearance of Glucosinolate Metabolites After Consumption of Cooked Broccoli. Front Nutr. 2020 Sep 24;7:575092. doi: 10.3389/fnut.2020.575092. eCollection 2020. PMID 33072799